CLINICAL TRIAL: NCT07046338
Title: Lentiviral Vector-modified Autologous Hematopoietic Stem Cells for Metachromatic Leukodystrophy (MLD)
Brief Title: Lentiviral Hematopoietic Stem Cell Gene Therapy for MLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-25001
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Metachromatic Leukodystrophy (MLD)
Keywords: Metachromatic leukodystrophy (MLD); Lentiviral vector; Hematopoietic stem cells
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentiviral TYF-ARSA modified autologous HSCs (Experimental): Autologous HSCs transduced with lentiviral TYF-ARSA vector carrying the functional gene.
  Interventions: Genetic: Lentiviral TYF-ARSA correction of patient's autologous HSCs

INTERVENTIONS:
Genetic: Lentiviral TYF-ARSA correction of patient's autologous HSCs — Infusion of lentiviral TYF-ARSA modified autologous HSCs at 1~10x10^6 gene-modified cells per kg body weight.

SUMMARY:
This is a Phase I/II clinical trial of gene therapy for treating Metachromatic leukodystrophy (MLD) using a safety and efficacy improved self-inactivating lentiviral vector TYF-ARSA to transduce patient-derived hematopoietic stem cells (HSCs), with the goal of achieving therapeutic gene correction through transplantation of genetically modified HSCs. The primary objectives are to evaluate the safety and efficacy of the gene therapy clinical protocol.

DETAILED DESCRIPTION:
Metachromatic leukodystrophy (MLD) is a rare lysosomal storage disease. This disease is an inherited single gene autosomal recessive defect. MLD is caused by a mutation in the ARSA gene encoding arylsulfatase A which leads to a deficiency in sulfatide degradation, resulting in its accumulation in oligodendrocytes, Schwann cells and neurons. A critical level of sulfatide storage can trigger demyelination, the hallmark of MLD, which results in multiple neurological symptoms. MLD has different onset ages including late infancy (1-2 years), adolescence (4 years-before sexual maturity) and adulthood (after sexual maturity). MLD patients are normally rescued by hematopoietic stem cell transplantation (HSCT) from a matched healthy donor. However, HSCT must be performed at a very early stage of the disease and carries a significant risk of graft-versus-host disease (GVHD), which restricts its therapeutic opportunities in MLD patients. This trial aims to treat MLD using an improved self-inactivating lentiviral vector (LV) carrying a functional ARSA gene to transduce patient-derived HSCs in culture, then delivering these genetically corrected HSCs carrying the normal ARSA gene to correct the genetic defect. The primary objectives are to evaluate the safety of the improved LV TYF-ARSA and the clinical protocol for gene therapy using the genetically modified HSCs, and the therapeutic efficacy in patients after treatment, assessment of vector integration sites, and finally the long-term correction of the pathological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 1 month
2. ARSA gene sequence analysis to confirm MLD mutations
3. Brain MR Imaging
4. Parent / guardian / patient signing informed consent
5. Patients and their families have a strong willingness to participate in clinical trials, are willing to bear all the consequences caused by the failure of the trial, and sign the informed consent

Exclusion Criteria:

1. HIV positive
2. Experiencing uncontrolled viral, bacterial or fungal infections, malignant tumors, heart abnormalities, liver dysfunction, or renal insufficiency
3. Cannot perform an MRI
4. Infection or dermatosis at infusion site
5. Any condition that may increase the subject's risk or interfere with the results of the trial, e.g. in addition to MLD, there are other neurological disorders.

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety of auto-HSCs transduced with lentiviral TYF-ARSA | up to 1 year follow up
  Safety of HSCs transduced with lentiviral TYF-ARSA, determined by number of participants with treatment-related adverse events (AEs), according to scheduled assessments, vital signs, & physical examinations as assessed by CTCAE v4.0. AEs & clinically significant abnormalities (meeting grade 3, 4, or 5 criteria according to CTCAE) will be summarized. AEs will be graded if related to the treatment.
Altered disease progression | up to 3 year follow up after treatment]
  Altered disease progression based on biochemical analysis.
Altered disease progression | up to 3 year follow up after treatment]
  Altered disease progression based on MRI brain imaging analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No